CLINICAL TRIAL: NCT00500929
Title: Mini-Metrxics: A Single-Centre, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Clinical Trial of CMI X-11S in Higher Risk Geriatric Patients Undergoing Open-Heart Surgical Procedures (OHSP)
Brief Title: A Clinical Trial in Higher Risk Geriatric Patients Undergoing OHSP
Acronym: MiniMetrxics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiometabolics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMI X-11S-G-1
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Heart Disease
Keywords: OHSP; High risk; Geriatrics
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CMI X-11S

SUMMARY:
To provide information on parameters needed to design a subsequent Phase III confirmatory trial and to assess the safety and efficacy of the acute use of CMI X-11S in high-risk geriatric patients undergoing open-heart surgical procedures (OHSP) requiring cardio-pulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Requirement for open-heart (including emergency) surgical procedures requiring cardio-pulmonary bypass:

  * Either:

    * Age ≥ 70 to <80 with a Parsonnet Mortality Risk Score of ≥13 (poor risk); OR
    * Age ≥ 80

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
ICU Time | 30 to 45 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shaohua Wang, Dr., Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada